CLINICAL TRIAL: NCT03004157
Title: A Randomized Comparison of Three Chest Compression Techniques and Associated Hemodynamic Effect During Infant CPR: a Randomized Manikin Study
Brief Title: Infant Chest Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Jacek Smereka (Unknown); Antonio Rodríguez-Núñez (Unknown); Jerzy R Ladny (Unknown); Steve Leung (Unknown); Kurt Ruetzler (Unknown)
Responsible Party: Principal Investigator, Łukasz Szarpak, PhD, DPH, EMT-P, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Infant11/2016
Record Dates: First submitted 2016-12-21; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Cardiopulmonary Arrest
Keywords: infant; cardiopulmonary resuscitation; hemodynamics; chest compressions
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Two finger technique (Experimental): Two finger technique TFT: the pediatric thorax is compressed with the tips of two fingers and is recommended for lone rescuer during infant CPR by international CPR guidelines
  Interventions: Procedure: cardiopulmonary resuscitation
- Two thumb technique (Experimental): Two thumb technique TTHT: the two thumbs of the rescuer are placed over the lower third of the sternum, with the fingers encircling the torso and supporting the back. This technique is recommended for two rescuers during infant CPR by international CPR guidelines
  Interventions: Procedure: cardiopulmonary resuscitation
- new two-thumb technique (Experimental): new two-thumb technique' (nTTT): this technique consists in using two thumbs directed at the angle of 90 degrees to the chest while closing the fingers of both hands in a fist
  Interventions: Procedure: cardiopulmonary resuscitation

INTERVENTIONS:
Procedure: cardiopulmonary resuscitation — CPR for 10 minutes with a chest compression: ventilation ratio of 15:2 according to international CPR guidelines

SUMMARY:
Pediatric cardiac arrest is an uncommon but critical life-threatening event requiring effective cardiopulmonary resuscitation (CPR). About 16,000 pediatric cardiac arrests occurs in the United States annually. Only 8% of the patients survive to hospital discharge and of these, up to two-thirds have neurological sequelae. Majority of pediatric cardiac arrest are below age of two and have poorer chance of survival versus older children

ELIGIBILITY:
Inclusion Criteria:

* active paramedics
* voluntary consent

Exclusion Criteria:

* pregnancy
* back pain
* wrist pain

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | 1 day
  The blood measurement system was calibrated before each CPR setting and blood pressure including systolic blood pressure (SBP)

SECONDARY OUTCOMES:
diastolic blood pressure | 1 day
  The blood measurement system was calibrated before each CPR setting and blood pressure including diastolic blood pressure (DBP)
mean arterial pressure | 1 day
  The blood measurement system was calibrated before each CPR setting and blood pressure including systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided